CLINICAL TRIAL: NCT04342052
Title: Glaucoma After Congenital Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: CCPMOH2020
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Glaucoma; Congenital Cataract
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the incidence of glaucoma following bilateral congenital cataract removal and estimate the associated risk factors in a large cohort to provide guidance for clinical practice.

DETAILED DESCRIPTION:
A prospective longitudinal cohort study of pediatric patients who underwent surgery for congenital/infantile cataracts between January 2011 and December 2025 was performed.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of bilateral congenital cataracts, the etiologies include congenital idiopathic cataract and congenital cataract associated with a systemic syndrome or ocular anomalies;
* cataract surgery performed in ZOC;
* age at cataract removal younger than 16 years;

Exclusion Criteria:

* the preoperative IOP was above 21 mm Hg;
* family history of glaucoma;
* signs of preoperative glaucoma were present, such as corneal clouding, corneal enlargement, excessive cup-disc ratio and myopic shift;
* ocular trauma history;
* previous surgery intervention and
* they were noncompliant with our follow-up protocol to monitor the occurrence of glaucoma and glaucoma suspect.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A prospective longitudinal cohort study of pediatric patients who underwent surgery for congenital cataracts was performed.
Sampling Method: Non-Probability Sample
Enrollment: 351 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of glaucoma after congenital cataract surgery | baseline
  A Kaplan-Meier analysis was used

SECONDARY OUTCOMES:
Risk factors of glaucoma after congenital cataract surgery | baseline
  Piecewise exponential survival models with mixed effects (PEWSMME) were used.(variables including demographic characters, surgery categories, clinical history, length of follow up).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Wu X, Wang Q, Zhou F, Chen H, Chen W, Lin D, Zhang X, Wang R, Chen J, Liu Z, Lin Z, Li X, Li J, Han Y, Liu Y, Lin H, Chen W. Incidence of and risk factors for suspected and definitive glaucoma after bilateral congenital cataract surgery: a 5-year follow-up. Br J Ophthalmol. 2024 Feb 21;108(3):476-483. doi: 10.1136/bjo-2022-322589. PMID 36828619